CLINICAL TRIAL: NCT02031276
Title: A Phase II, Multicenter, Randomized, Double-blind, Multiple Dose, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy, Pharmacokinetics, and Safety of BI 655066/ABBV-066 (Risankizumab), an IL-23 p19 Antagonist Monoclonal Antibody, in Patients With Moderately to Severely Active Crohn's Disease, Who Are naïve to, or Were Previously Treated With Anti-TNF Therapy
Brief Title: Efficacy, Safety and Pharmacokinetics of BI 655066/ABBV-066 (Risankizumab) in Patients With Active, Moderate-to-severe Crohn's Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M15-993; 2013-002902-29 (EudraCT Number); 1311.6 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2013-12-16; First posted 2014-01-09 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-10

CONDITIONS: Crohn Disease
Keywords: ABBV-066; BI 655066; risankizumab
MeSH Terms: conditions — Crohn Disease | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Period 1 was blinded intravenous (IV) therapy, period 2 was open label IV therapy and period 3 was open label subcutaneous (SC) therapy.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Double-blind Placebo IV (Placebo Comparator): Participants randomized to receive double-blind placebo for risankizumab by intravenous (IV) injection for 12 weeks in Period 1, followed by open-label risankizumab 600 mg IV in Period 2, then open-label risankizumab 180 mg by subcutaneous (SC) injection in Period 3.
  Interventions: Drug: risankizumab IV; Drug: risankizumab SC; Drug: Placebo
- Double-blind Risankizumab 200 mg IV (Experimental): Participants randomized to receive double-blind risankizumab 200 mg by intravenous (IV) injection for 12 weeks in Period 1, followed by open-label risankizumab 600 mg IV in Period 2, then open-label risankizumab 180 mg by subcutaneous (SC) injection in Period 3.
  Interventions: Drug: risankizumab IV; Drug: risankizumab SC
- Double-blind Risankizumab 600 mg IV (Experimental): Participants randomized to receive double-blind risankizumab 600 mg by intravenous (IV) injection for 12 weeks in Period 1, followed by open-label risankizumab 600 mg IV in Period 2, then open-label risankizumab 180 mg by subcutaneous (SC) injection in Period 3.
  Interventions: Drug: risankizumab IV; Drug: risankizumab SC

INTERVENTIONS:
Drug: risankizumab IV — risankizumab administered by IV infusion
  Other Names: BI 655066; ABBV-066
Drug: risankizumab SC — risankizumab administered by SC injection
  Other Names: BI 655066; ABBV-066
Drug: Placebo — Placebo for risankizumab administered by IV infusion
  Arms: Double-blind Placebo IV

SUMMARY:
This study is a proof of concept, multi-center, randomized, double-blind, placebo-controlled, parallel-group phase 2 dose-ranging study of BI 655066/ABBV-066 (risankizumab), an IL-23 p19 antagonist monoclonal antibody, in patients with moderately to severely active Crohn's disease.

ELIGIBILITY:
Inclusion criteria:

1. Men or women 18-75 years at the time of consent.
2. Diagnosis of Crohn's disease (CD) at least 3 months prior to screening.
3. Moderate to severe active CD, defined as Crohn's Disease Activity Index (CDAI) ≥ 220 and ≤ 450.
4. Presence of mucosal ulcers in at least one segment of the ileum or colon and a Crohn's Disease Endoscopic Index of Severity (CDEIS) score ≥ 7 (for patients with isolated ileitis, ≥4), as assessed by ileocolonoscopy and confirmed by central independent reviewer before randomization
5. Patients who are naive or experienced to 1 or more TNF antagonists (infliximab, adalimumab, or certolizumab pegol) at a dose approved for CD. TNF antagonist experienced patients may have stopped anti-TNF treatment due to primary or secondary non-responsiveness, intolerance or for other reasons.
6. Female patients:

   Women of childbearing potential (not surgically sterilized and between menarche and 1 year postmenopause), that, if sexually active agree to use one of the appropriate medically accepted methods of birth control in addition to the consistent and correct use of a condom from date of screening until 15 weeks after last administration of study medication. Medically accepted methods of contraception are: ethinyl estradiol containing contraceptives, diaphragm with spermicide substance, and intra-uterine-device, or
   1. Surgically sterilized female patients with documentation of prior hysterectomy, tubal ligation or complete bilateral oophorectomy, or
   2. Postmenopausal women with postmenopausal is defined as permanent cessation = 1 year of previously occurring menses, and
   3. Negative serum ß-Human Chorionic Gonadotrophin (ß-HCG) test at screening and urine pregnancy test prior to randomization.

   Male patients:
   1. Who are documented to be sterile, or
   2. Who consistently and correctly use effective method of contraception (i.e. condoms) during the study and 15 weeks after last administration of study medication.
7. Have the capacity to understand and sign an informed consent form.
8. Be able to adhere to the study visit schedule and other protocol requirements.

Exclusion criteria:

1. Have complications of CD such as strictures, stenoses, short gut syndrome, or any other manifestation that might require surgery, could preclude the use of the CDAI to assess response to therapy, or would possibly confound the evaluation of benefit from treatment with BI 655066.
2. Have any current or prior abscesses, unless they have been drained and treated at least 6 weeks prior to randomization and are not anticipated to require surgery. Patients with active fistulas may be included if there is no anticipation of a need for surgery and there are currently no abscesses present.
3. Have had any kind of bowel resection or diversion within 6 months or any other intra-abdominal surgery within 3 months prior to screening. Patients with a current ileostomy or colostomy are excluded.
4. Have received treatment with:

   * Total parenteral nutrition (TPN) within 2 weeks of screening.
   * Any dose of ustekinumab (Stelara®).
   * Anti-TNF therapy ≤ 8 weeks prior to the first administration of study medication or any other biologic ≤ 8 weeks prior to the first administration of study drug or within 5 times the half-life of the biologic prior to the first administration of study agent, whichever is longer.
   * Natalizumab, efalizumab, or agents that deplete B or T cells (e.g., rituximab, alemtuzumab, or visilizumab) within 6 months of screening, or, if after receiving these agents, evidence is available at screening of persistent depletion of the targeted lymphocyte population.
   * Any investigational drug within the previous 4 weeks or 5 times the half-life of the investigational agent prior to the first administration of study agent, whichever is longer.
   * Regular daily use of opioids for medical reasons within previous 3 months prior to the first administration of study agent.
   * Rectal 5-aminosalicylic acid (5-ASA) compounds, parenteral or rectal corticosteroids must have been discontinued at least 4 weeks prior to visit 2.
   * Cannot adhere to the concomitant medication requirements specified in section 4.2.2.
5. Are pregnant, nursing, or planning pregnancy (both men and women) while enrolled in the study, or within 15 weeks after receiving the last dose of study medication.
6. Have used apheresis (e.g., Adacolumn apheresis) ≤ 2 weeks prior to screening.
7. Have received any live bacterial or viral vaccination ≤ 12 weeks prior to Day 1. Patients must agree not to receive a live virus or bacterial vaccination during the study or up to 12 months after the last administration of study drug.
8. Have had a Bacille Calmette-Guérin (BCG) vaccination within 12 months of screening. Patient must agree not to receive a BCG vaccination during the study or up to 12 months after the last study drug administration.
9. Have signs or symptoms of infection, history of chronic or recurrent infection, have evidence of active herpes zoster infection ≤ 8 weeks of screening, have a stool culture or other examination positive for an enteric pathogen, have a history of latent or active granulomatous infection, infected with human immunodeficiency virus (HIV), hepatitis B (HepB) or hepatitis C (HepC) virus, established nonserious infections
10. Are not eligible according to tuberculosis (TB) screening criteria
11. Have severe, progressive or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac, neurologic, cerebral or psychiatric disease or signs and symptoms.
12. Have a transplanted organ
13. Have known history of lymphoproliferative disease
14. Have any malignancy or history of malignancy
15. Have previously undergone allergy immunotherapy
16. Are unable or unwilling to undergo multiple venipunctures
17. Are known to have substance abuse
18. Are currently or intending to participate in any other study
19. Have screening laboratory test results within the protocol stated parameters
20. Have a known hypersensitivity to study drug
21. Have evidence of current or previous clinically significant disease, medical condition other than CD, finding of the medical examination or lab value.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

REFERENCES:
- [Derived] Feagan BG, Panes J, Ferrante M, Kaser A, D'Haens GR, Sandborn WJ, Louis E, Neurath MF, Franchimont D, Dewit O, Seidler U, Kim KJ, Selinger C, Padula SJ, Herichova I, Robinson AM, Wallace K, Zhao J, Minocha M, Othman AA, Soaita A, Visvanathan S, Hall DB, Bocher WO. Risankizumab in patients with moderate to severe Crohn's disease: an open-label extension study. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):671-680. doi: 10.1016/S2468-1253(18)30233-4. Epub 2018 Jul 25. PMID 30056030
- [Derived] Feagan BG, Sandborn WJ, D'Haens G, Panes J, Kaser A, Ferrante M, Louis E, Franchimont D, Dewit O, Seidler U, Kim KJ, Neurath MF, Schreiber S, Scholl P, Pamulapati C, Lalovic B, Visvanathan S, Padula SJ, Herichova I, Soaita A, Hall DB, Bocher WO. Induction therapy with the selective interleukin-23 inhibitor risankizumab in patients with moderate-to-severe Crohn's disease: a randomised, double-blind, placebo-controlled phase 2 study. Lancet. 2017 Apr 29;389(10080):1699-1709. doi: 10.1016/S0140-6736(17)30570-6. Epub 2017 Apr 12. PMID 28411872

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 1 of 3 double-blind treatment arms in Period 1; those who achieved deep remission in Period 1 entered Period 2 washout; those who did not achieve deep remission in Period 1 entered Period 2 open-label (OL) treatment. Participants who were in clinical remission at the end of Period 2 continued to Period 3 OL treatment
Period: Period 1 Double-blind IV
Arm/Group | Double-blind Placebo IV | Double-blind Risankizumab 200 mg IV | Double-blind Risankizumab 600 mg IV
Started | 39 | 41 | 41
Completed | 33 | 35 | 40
Not Completed | 6 | 6 | 1
Not completed — Adverse Event | 6 | 5 | 1
Not completed — Other | 0 | 1 | 0
Period: Period 2 Open-label Risankizumab IV
Arm/Group | Double-blind Placebo IV | Double-blind Risankizumab 200 mg IV | Double-blind Risankizumab 600 mg IV
Started | 33 | 35 | 39 (1 participant did not enter Period 2 (declined open-label treatment in Period 2))
Completed | 29 | 33 | 38
Not Completed | 4 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Other | 0 | 2 | 1
Period: Period 3 Open-label Risankizumab SC
Arm/Group | Double-blind Placebo IV | Double-blind Risankizumab 200 mg IV | Double-blind Risankizumab 600 mg IV
Started | 19 (10 participants did not enter period 3 (not in clinical remission)) | 22 (11 participants did not enter period 3 (not in clinical remission)) | 21 (17 participants did not enter period 3 (not in clinical remission))
Completed | 16 | 19 | 19
Not Completed | 3 | 3 | 2
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set - Period 1 (FAS-P1): All randomized subjects who received at least 1 dose of study drug in the double-blind IV period (Period 1).
Groups:
- Double-blind Placebo IV: Participants randomized in Period 1 to receive double-blind placebo for risankizumab by intravenous (IV) injection for 12 weeks in Period 1, followed by open-label risankizumab 600 mg IV in Period 2, then open-label risankizumab 180 mg by subcutaneous (SC) injection in Period 3.
- Double-blind Risankizumab 200 mg IV: Participants randomized in Period 1 to receive double-blind risankizumab 200 mg by intravenous (IV) injection for 12 weeks in Period 1, followed by open-label risankizumab 600 mg IV in Period 2, then open-label risankizumab 180 mg by subcutaneous (SC) injection in Period 3.
- Double-blind Risankizumab 600 mg IV: Participants randomized in Period 1 to receive double-blind risankizumab 600 mg by intravenous (IV) injection for 12 weeks in Period 1, followed by open-label risankizumab 600 mg IV in Period 2, then open-label risankizumab 180 mg by subcutaneous (SC) injection in Period 3.
- Total: Total of all reporting groups
Arm/Group | Double-blind Placebo IV | Double-blind Risankizumab 200 mg IV | Double-blind Risankizumab 600 mg IV | Total
Number analyzed (Participants) | 39 | 41 | 41 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (13.86) | 38.8 (13.27) | 39.9 (13.26) | 38.1 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 16 | 47
  Male | 23 | 26 | 25 | 74

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Disease Activity Index (CDAI) Clinical Remission at Week 12
Description: The CDAI is a measure of clinical response and remission. The CDAI includes 8 variables encompassing both patient-reported (symptoms, general well-being) and objective (medication usage, laboratory variables, presence of abdominal mass or complications, and weight) variables. For symptoms scores, patients keep track of daily symptoms on a diary card and the daily symptom scores are summed for the week. Each item in the CDAI is assigned a specific weight, and the weighted values of the items are totaled to produce the CDAI. Higher CDAI scores indicate greater disease activity, with a lower limit of 0 and no set upper limit: < 150 indicates remission, 150 - 219 indicates mildly active disease, 220 - 450 indicates moderately active disease, and > 450 indicates severely active disease. CDAI clinical remission is defined as CDAI < 150 at Week 12. Nonresponder imputation (NRI): missing values were counted as nonresponders.
Time Frame: Week 12
Population: Full Analysis Set-Period 1 (FAS-P1): All randomized subjects who received at least 1 dose of study drug in the double-blind IV period (Period 1).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Double-blind Placebo IV (Period 1): Participants randomized to receive double-blind placebo for risankizumab by intravenous (IV) injection for 12 weeks.
- Double-blind Risankizumab 200 mg IV (Period 1): Participants randomized to receive double-blind risankizumab 200 mg by intravenous (IV) injection for 12 weeks.
- Double-blind Risankizumab 600 mg IV (Period 1): Participants randomized to receive double-blind risankizumab 600 mg by intravenous (IV) injection for 12 weeks.
- Double-blind Risankizumab 200 + 600 mg IV (Period 1): Participants randomized to receive double-blind risankizumab 200 mg and 600 mg by intravenous (IV) injection for 12 weeks.
Arm/Group | Double-blind Placebo IV (Period 1) | Double-blind Risankizumab 200 mg IV (Period 1) | Double-blind Risankizumab 600 mg IV (Period 1) | Double-blind Risankizumab 200 + 600 mg IV (Period 1)
Number analyzed (Participants) | 39 | 41 | 41 | 82
percentage of participants | 15.4 [5.9 to 30.5] | 19.5 [8.8 to 34.9] | 36.6 [22.1 to 53.1] | 28.0 [18.7 to 39.1]
Statistical Analysis 1: Comparison: Double-blind Placebo IV (Period 1) vs Double-blind Risankizumab 200 + 600 mg IV (Period 1); Statistics for the difference are calculated using the Cochran-Mantel-Haenszel risk difference stratified by anti-tumor necrosis factor (anti-TNF) exposure; Test type: Other; p = 0.0955, Cochran-Mantel-Haenszel; difference in percentage of participants = 12.6, 95% CI 2-sided [-2.2 to 27.5]

2. Secondary Outcome: Percentage of Participants Achieving CDAI Clinical Response at Week 12
Description: The CDAI is a measure of clinical response and remission. The CDAI includes 8 variables encompassing both patient-reported (symptoms, general well-being) and objective (medication usage, laboratory variables, presence of abdominal mass or complications, and weight) variables. For symptoms scores, patients keep track of daily symptoms on a diary card and the daily symptom scores are summed for the week. Each item in the CDAI is assigned a specific weight, and the weighted values of the items are totaled to produce the CDAI. Higher CDAI scores indicate greater disease activity, with a lower limit of 0 and no set upper limit: < 150 indicates remission, 150 - 219 indicates mildly active disease, 220 - 450 indicates moderately active disease, and > 450 indicates severely active disease. CDAI clinical response is defined as either a CDAI < 150 or a CDAI reduction from Baseline of at least 100 points at Week 12. NRI: missing values were counted as nonresponders.
Time Frame: Week 12
Population: FAS-P1: All randomized subjects who received at least 1 dose of study drug in the double-blind IV period (Period 1).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind Placebo IV (Period 1) | Double-blind Risankizumab 200 mg IV (Period 1) | Double-blind Risankizumab 600 mg IV (Period 1) | Double-blind Risankizumab 200 + 600 mg IV (Period 1)
Number analyzed (Participants) | 39 | 41 | 41 | 82
percentage of participants | 23.1 [11.1 to 39.3] | 31.7 [18.1 to 48.1] | 41.5 [26.3 to 57.9] | 36.6 [26.2 to 48.0]
Statistical Analysis 1: Comparison: Double-blind Placebo IV (Period 1) vs Double-blind Risankizumab 200 + 600 mg IV (Period 1); Statistics for the difference are calculated using the Cochran-Mantel-Haenszel risk difference stratified by anti-TNF exposure; Test type: Other; p = 0.1151, Cochran-Mantel-Haenszel; difference in percentage of participants = 13.4, 95% CI 2-sided [-3.3 to 30.1]

3. Secondary Outcome: Percentage of Participants Achieving Crohn's Disease Endoscopic Index of Severity (CDEIS) Remission at Week 12
Description: CDEIS is an index for determining the severity of Crohn's disease with endoscopic localization to ileum and colon. CDEIS considers 4 parameters (deep ulcerations, superficial ulcerations, surface involved by disease, and surface involved by ulcerations), each one evaluated in 5 pre-defined segments of the colon (ileum, ascending colon, transverse colon, descending colon and sigmoid loop, and rectum). The results of the individual segments of the colon are divided by the number of segments investigated; the presence of stenosis increases the score at the end of the computation. CDEIS remission is defined as a CDEIS ≤ 4 (or, for patients with initial isolated ileitis, a CDEIS ≤ 2) at Week 12. NRI: missing values were counted as nonresponders.
Time Frame: Week 12
Population: FAS-P1: All randomized subjects who received at least 1 dose of study drug in the double-blind IV period (Period 1).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind Placebo IV (Period 1) | Double-blind Risankizumab 200 mg IV (Period 1) | Double-blind Risankizumab 600 mg IV (Period 1) | Double-blind Risankizumab 200 + 600 mg IV (Period 1)
Number analyzed (Participants) | 39 | 41 | 41 | 82
percentage of participants | 2.6 [0.1 to 13.5] | 9.8 [2.7 to 23.1] | 19.5 [8.8 to 34.9] | 14.6 [7.8 to 24.2]
Statistical Analysis 1: Comparison: Double-blind Placebo IV (Period 1) vs Double-blind Risankizumab 200 + 600 mg IV (Period 1); [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0057, Cochran-Mantel-Haenszel; difference in percentage of participants = 12.0, 95% CI 2-sided [3.5 to 20.6]

4. Secondary Outcome: Percentage of Participants Achieving CDEIS Response at Week 12
Description: CDEIS is an index for determining the severity of Crohn's disease with endoscopic localization to ileum and colon. CDEIS considers 4 parameters (deep ulcerations, superficial ulcerations, surface involved by disease, and surface involved by ulcerations), each one evaluated in 5 pre-defined segments of the colon (ileum, ascending colon, transverse colon, descending colon and sigmoid loop, and rectum). The results of the individual segments of the colon are divided by the number of segments investigated; the presence of stenosis increases the score at the end of the computation. CDEIS response is defined as defined as ≥ 50% reduction of CDEIS from Baseline to Week 12. NRI: missing values were counted as nonresponders.
Time Frame: Week 12
Population: FAS-P1: All randomized subjects who received at least 1 dose of study drug in the double-blind IV period (Period 1).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind Placebo IV (Period 1) | Double-blind Risankizumab 200 mg IV (Period 1) | Double-blind Risankizumab 600 mg IV (Period 1) | Double-blind Risankizumab 200 + 600 mg IV (Period 1)
Number analyzed (Participants) | 39 | 41 | 41 | 82
percentage of participants | 12.8 [4.3 to 27.4] | 26.8 [14.2 to 42.9] | 36.6 [22.1 to 53.1] | 31.7 [21.9 to 42.9]
Statistical Analysis 1: Comparison: Double-blind Placebo IV (Period 1) vs Double-blind Risankizumab 200 + 600 mg IV (Period 1); [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0104, Cochran-Mantel-Haenszel; difference in percentage of participants = 18.7, 95% CI 2-sided [4.4 to 33.0]

5. Secondary Outcome: Percentage of Participants Achieving Mucosal Healing at Week 12
Description: Mucosal healing was defined as the absence of mucosal ulceration, i.e., a CDEIS ulceration sub-score (deep ulceration, superficial ulceration, ulcerated stenosis) of 0 at Week 12. NRI: missing values were counted as nonresponders.
Time Frame: Week 12
Population: FAS-P1: All randomized subjects who received at least 1 dose of study drug in the double-blind IV period (Period 1).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind Placebo IV (Period 1) | Double-blind Risankizumab 200 mg IV (Period 1) | Double-blind Risankizumab 600 mg IV (Period 1) | Double-blind Risankizumab 200 + 600 mg IV (Period 1)
Number analyzed (Participants) | 39 | 41 | 41 | 82
percentage of participants | 2.6 [0.1 to 13.5] | 2.4 [0.1 to 12.9] | 7.3 [1.5 to 19.9] | 4.9 [1.3 to 12.0]
Statistical Analysis 1: Comparison: Double-blind Placebo IV (Period 1) vs Double-blind Risankizumab 200 + 600 mg IV (Period 1); [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.4977, Cochran-Mantel-Haenszel; difference in percentage of participants = 2.4, 95% CI 2-sided [-4.5 to 9.2]

6. Secondary Outcome: Percentage of Participants Achieving Deep Remission at Week 12
Description: Deep remission is defined as clinical remission (CDAI < 150) AND CDEIS remission (CDEIS ≤ 4, or ≤ 2 in participants with initial isolated ileitis) at Week 12. NRI: missing values were counted as nonresponders.
Time Frame: Week 12
Population: FAS-P1: All randomized subjects who received at least 1 dose of study drug in the double-blind IV period (Period 1).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind Placebo IV (Period 1) | Double-blind Risankizumab 200 mg IV (Period 1) | Double-blind Risankizumab 600 mg IV (Period 1) | Double-blind Risankizumab 200 + 600 mg IV (Period 1)
Number analyzed (Participants) | 39 | 41 | 41 | 82
percentage of participants | 0 [0.0 to 9.0] | 2.4 [0.1 to 12.9] | 12.2 [4.1 to 26.2] | 7.3 [2.7 to 15.2]
Statistical Analysis 1: Comparison: Double-blind Placebo IV (Period 1) vs Double-blind Risankizumab 200 + 600 mg IV (Period 1); [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0107, Cochran-Mantel-Haenszel; difference in percentage of participants = 7.4, 95% CI 2-sided [1.7 to 13.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 15 weeks after the last dose of study drug (up to 67 weeks).
Description: TEAEs and TESAEs: AEs and SAEs with onset/worsening from the first dose of DB study drug until either the first dose of open-label (OL) risankizumab or 15 weeks after the last dose of DB study drug (up to 27 weeks); for All Risankizumab, from the first dose of DB or OL risankizumab until 15 weeks after the last dose of risankizumab (up to 67 weeks).
Groups:
- Double-blind Placebo IV (Period 1): Participants received double-blind placebo for risankizumab by intravenous (IV) injection for 12 weeks.
- Double-blind Risankizumab 200 mg IV (Period 1): Participants received double-blind risankizumab 200 mg by intravenous (IV) injection for 12 weeks.
- Double-blind Risankizumab 600 mg IV (Period 1): Participants administered double-blind risankizumab 600 mg by intravenous (IV) injection for 12 weeks.
- Open-label Risankizumab 600 mg IV (Period 2): Participants administered open-label risankizumab 600 mg by intravenous (IV) injection for 12 weeks.
- Open-label Risankizumab 180 mg SC (Period 3): Participants administered open-label risankizumab 600 mg by subcutaneous (SC) injection for 12 weeks.
- All Risankizumab: Participants administered at least one dose of risankizumab.
Arm/Group | Double-blind Placebo IV (Period 1) | Double-blind Risankizumab 200 mg IV (Period 1) | Double-blind Risankizumab 600 mg IV (Period 1) | Open-label Risankizumab 600 mg IV (Period 2) | Open-label Risankizumab 180 mg SC (Period 3) | All Risankizumab
Serious Adverse Events (participants affected / at risk) | 13/39 | 10/41 | 4/41 | 11/101 | 7/62 | 31/115
Other Adverse Events (participants affected / at risk) | 28/39 | 25/41 | 21/41 | 48/101 | 31/62 | 80/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo IV (Period 1) (N=39) | Double-blind Risankizumab 200 mg IV (Period 1) (N=41) | Double-blind Risankizumab 600 mg IV (Period 1) (N=41) | Open-label Risankizumab 600 mg IV (Period 2) (N=101) | Open-label Risankizumab 180 mg SC (Period 3) (N=62) | All Risankizumab (N=115)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1
BLINDNESS TRANSIENT (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
DIPLOPIA (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
ANAL FISTULA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
APHTHOUS ULCER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 5 | 2 | 1 | 3 | 1 | 7
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 3
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 2
PROCTALGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 3
ASTHENIA (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
PAIN (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
PYREXIA (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
ABDOMINAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1
APPENDICITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
INCISION SITE ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
OSTEOMYELITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1
RECTAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
VAGINAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
BLOOD MAGNESIUM DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 2
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
CEREBROSPINAL FLUID LEAKAGE (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
HEMIPARESIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
MIGRAINE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
PSYCHIATRIC DECOMPENSATION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
ABORTION INDUCED (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo IV (Period 1) (N=39) | Double-blind Risankizumab 200 mg IV (Period 1) (N=41) | Double-blind Risankizumab 600 mg IV (Period 1) (N=41) | Open-label Risankizumab 600 mg IV (Period 2) (N=101) | Open-label Risankizumab 180 mg SC (Period 3) (N=62) | All Risankizumab (N=115)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 3 | 2 | 1 | 6
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 6 | 4 | 11 | 5 | 21
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2 | 1 | 2 | 3 | 8
CROHN'S DISEASE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 4 | 4
DIARRHOEA (Gastrointestinal disorders) | 2 | 2 | 3 | 4 | 1 | 9
HAEMATOCHEZIA (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 1 | 4
NAUSEA (Gastrointestinal disorders) | 4 | 9 | 4 | 6 | 1 | 18
VOMITING (Gastrointestinal disorders) | 4 | 4 | 2 | 7 | 0 | 11
ASTHENIA (General disorders) | 2 | 4 | 2 | 3 | 1 | 9
FATIGUE (General disorders) | 3 | 0 | 2 | 2 | 5 | 8
INFLUENZA LIKE ILLNESS (General disorders) | 2 | 1 | 2 | 0 | 0 | 3
MALAISE (General disorders) | 0 | 0 | 1 | 4 | 2 | 7
PERIPHERAL SWELLING (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 3 | 3 | 3 | 6 | 3 | 14
NASOPHARYNGITIS (Infections and infestations) | 3 | 2 | 2 | 8 | 9 | 18
SINUSITIS (Infections and infestations) | 0 | 1 | 1 | 2 | 3 | 7
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3 | 0 | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 1 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 | 0 | 1 | 2 | 0 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 6 | 8 | 7 | 6 | 25
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 3 | 2 | 9
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 0 | 4
DIZZINESS (Nervous system disorders) | 1 | 1 | 3 | 5 | 1 | 9
HEADACHE (Nervous system disorders) | 5 | 6 | 5 | 7 | 6 | 22
LETHARGY (Nervous system disorders) | 3 | 0 | 0 | 2 | 1 | 2
INSOMNIA (Psychiatric disorders) | 0 | 1 | 3 | 1 | 2 | 6
SLEEP DISORDER (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 3 | 3 | 7
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 4 | 2 | 8
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 3 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.